CLINICAL TRIAL: NCT03377244
Title: Healthy Body Healthy Souls: A Weight Loss Intervention Using Diabetes Prevention Program Lifestyle Intervention (DPP-LI) With Church Level Systems Change in the Marshallese Population
Brief Title: Healthy Body Healthy Souls in the Marshallese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 217566
Record Dates: First submitted 2017-12-07; First posted 2017-12-19 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Weight Loss; Pre Diabetes; Overweight and Obesity
Keywords: Marshallese; Pacific Islanders
MeSH Terms: conditions — Weight Loss; Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Our aim is to pilot test a multi-level weight-loss intervention in the Marshallese community. Changes in outcomes were examined from baseline to 6 months post-intervention (12 months post-initiation of the intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBHS (Experimental): Participants in the Healthy Bodies Healthy Souls (HBHS) arm received the Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program Lifestyle Intervention (WORD DPP) with the addition of church-level policy changes to support the individual behavioral intervention of the WORD DPP. The WORD DPP is a faith-based diabetes prevention curriculum that teaches participants to connect faith and health to have a healthy weight, eat healthy, and be physically active. The WORD DPP includes 16 modules that are intended to be delivered over a 24 week period, each module approximately 90 minutes in length. Church-level changes to support healthier behaviors include improvements in food purchasing and preparation for events, physical activity programs, and increased congregational engagement in health promotion activities.
  Interventions: Behavioral: HBHS
- HBHS Policy (Active Comparator): Participants in the HBHS Policy arm included members of churches enrolled in the HBHS study who did not receive the WORD DPP intervention (ie, these participants were exposed to only the church-level policy changes). Church-level changes to support healthier behaviors include improvements in food purchasing and preparation for events, physical activity programs, and increased congregational engagement in health promotion activities.
  Interventions: Behavioral: HBHS Policy
- WORD DPP (Other): Participants in the Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program Lifestyle Intervention (WORD DPP) arm included participants enrolled in a separate DPP study without the church-level policy changes (ie, these participants received only the WORD DPP intervention). The WORD DPP is a faith-based diabetes prevention curriculum that teaches participants to connect faith and health to have a healthy weight, eat healthy, and be physically active. The WORD DPP-LI includes 16 modules that are intended to be delivered over a 24 week period, each module approximately 90 minutes in length.
  Interventions: Behavioral: WORD DPP

INTERVENTIONS:
Behavioral: HBHS — Faith based diabetes curriculum that teaches participants to connect faith and health plus church-level policy changes that encourages participants to engage in healthy behaviors.
  Arms: HBHS
Behavioral: HBHS Policy — Church-level policy changes that encourages participants to engage in healthy behaviors.
  Arms: HBHS Policy
Behavioral: WORD DPP — Faith based diabetes curriculum that teaches participants to connect faith and health.
  Arms: WORD DPP

SUMMARY:
The primary aim is to pilot test a weight-loss intervention for Marshallese adults, referred to throughout as Healthy Bodies Healthy Souls (HBHS). The HBHS intervention includes the Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program Lifestyle Intervention (WORD DPP) implemented at the individual level, with the additional enhancement of working with Marshallese churches to implement church-level changes to support the individual behavioral intervention of the WORD DPP. We will then compare changes in outcomes with participants in the churches who were exposed to the policy changes but did not participate in the WORD DPP, and with those enrolled in a separate DPP trial who participated in the WORD DPP but were not exposed to church-level policy changes.

DETAILED DESCRIPTION:
Background and Rationale

Disparities in type 2 diabetes, pre-diabetes, and obesity among the Marshallese and Pacific Islanders.

This study focuses on the Marshallese living in Arkansas. The Marshallese are a Pacific Islander population experiencing significant health disparities, with some of the highest documented rates of type 2 diabetes of any population group in the world. Our review of local, national, and international data sources found estimates of diabetes in the Marshallese population (in the US and the Republic of the Marshall Islands) ranging from 20% to 50%, compared to 8% for the US population and 4% worldwide.

While national prevalence data are limited, 23.7% of Pacific Islanders surveyed by the Centers for Disease Control and Prevention (CDC) in 2010 reported a diagnosis of type 2 diabetes - more than all other racial/ethnic groups. Our preliminary research, which included health screenings with the Marshallese community in Northwest Arkansas (n = 401), documented extremely high incidence of diabetes (38.2%) and pre-diabetes (32.4%). Our pilot data also revealed similar disparities in obesity, one of the strongest risk factors for diabetes; 90% of Marshallese participants were classified as overweight or obese. Further compounding these significant disparities, Pacific Islanders living in the US are less likely than other racial/ethnic groups to receive preventive or diagnostic treatment or diabetes education.

This study addresses an urgent need for interventions to reduce obesity and diabetes disparities in the Marshallese community and will employ a culturally appropriate, multilevel approach. The scientific premise of our study includes four main points. First, the Marshallese in Arkansas suffer from a significant and disproportionate burden of type 2 diabetes and lack access to effective prevention and treatment due to a dearth of research with Pacific Islanders.Second, the association between weight gain and risk for type 2 diabetes is strong. Overweight/obesity is considered the strongest modifiable risk factor for type 2 diabetes, and even a modest reduction in weight (5-10%) is clinically meaningful. Third, research demonstrates the effectiveness of multi-level lifestyle interventions in reducing weight and the onset and impact of diabetes. Fourth, to be effective among Pacific Islanders, interventions must be developed to address influences at multiple levels and should be culturally adapted to incorporate Pacific Islanders' worldviews and cultural values. Prior research indicates the importance of using a Community Based Participatory Research (CBPR) approach to understand and integrate cultural nuances during the cultural adaptation process and implementation of multilevel interventions. A CBPR approach is also essential to conducting ethical, valid health research in populations whose health beliefs and behaviors have been shaped by historical trauma. Finally, churches are primary social institutions of Pacific Islander health. Faith-based interventions are effective at improving behavioral and anthropometric outcomes within collectivistic communities and therefore hold great promise for Marshallese and other Pacific Islanders.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported Marshallese
2. 18 years of age or older
3. To participate in the DPP-LI, have a body mass index (BMI) of ≥25 kg/m^2

Exclusion Criteria:

1. A clinically significant medical condition likely to impact weight (cancer, HIV/AIDS, etc.)
2. Currently pregnant or breastfeeding an infant who is 6 months old or younger.
3. Have any condition that makes it unlikely that the participant will be able to follow the protocol, such as terminal illness, plans to move out of the area within 6 months, and inability to finish the intervention, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pearl McElfish, PhD, MBA, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shannon J, Kristal AR, Curry SJ, Beresford SA. Application of a behavioral approach to measuring dietary change: the fat- and fiber-related diet behavior questionnaire. Cancer Epidemiol Biomarkers Prev. 1997 May;6(5):355-61. PMID 9149896
- [Background] Gruber KJ. Social support for exercise and dietary habits among college students. Adolescence. 2008 Fall;43(171):557-75. PMID 19086670
- [Background] Clark MM, Abrams DB, Niaura RS, Eaton CA, Rossi JS. Self-efficacy in weight management. J Consult Clin Psychol. 1991 Oct;59(5):739-44. doi: 10.1037//0022-006x.59.5.739. PMID 1955608
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Resnick B, Luisi D, Vogel A, Junaleepa P. Reliability and validity of the self-efficacy for exercise and outcome expectations for exercise scales with minority older adults. J Nurs Meas. 2004 Winter;12(3):235-47. doi: 10.1891/jnum.12.3.235. PMID 16138727
- See also: DASH 2 Brief Physical Activity Questionnaire (p. 116) — https://biolincc.nhlbi.nih.gov/media/studies/dashsodium/Forms_Manual.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- HBHS: Participants in the HBHS arm received the Wholeness, Oneness, Righteousness, Deliverance Diabetes Prevention Program Lifestyle Intervention (WORD DPP) with the addition of church-level policy changes to support the individual behavioral intervention of the WORD DPP. The WORD DPP is a faith-based diabetes prevention curriculum that teaches participants to connect faith and health to have a healthy weight, eat healthy, and be physically active. The WORD DPP-LI includes 16 modules that are intended to be delivered over a 24 week period, each module approximately 90 minutes in length. Church-level changes to support healthier behaviors include improvements in food purchasing and preparation for events, physical activity programs, and increased congregational engagement in health promotion activities.
  HBHS: Faith based diabetes curriculum that teaches participants to connect faith and health plus church-level policy changes that encourages participants to engage in healthy behaviors.
- WORD DPP: Participants in the WORD DPP arm included participants enrolled in a separate DPP study without the church-level policy changes (ie, these participants received only the WORD DPP intervention). The WORD DPP is a faith-based diabetes prevention curriculum that teaches participants to connect faith and health to have a healthy weight, eat healthy, and be physically active. The WORD DPP-LI includes 16 modules that are intended to be delivered over a 24 week period, each module approximately 90 minutes in length.
  WORD DPP: Faith based diabetes curriculum that teaches participants to connect faith and health.
Period: Baseline
Arm/Group | HBHS | HBHS Policy | WORD DPP
Started | 19 | 14 | 69
Completed | 19 | 14 | 69
Not Completed | 0 | 0 | 0
Period: 6 Months Post-intervention
Arm/Group | HBHS | HBHS Policy | WORD DPP
Started | 19 | 14 | 69
Completed | 13 | 7 | 55
Not Completed | 6 | 7 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HBHS | HBHS Policy | WORD DPP | Total
Number analyzed (Participants) | 19 | 14 | 69 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (9.8) | 27.3 (8.4) | 43.7 (9.8) | 40.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 44 | 63
  Male | 8 | 6 | 25 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 19 | 14 | 69 | 102
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 14 | 69 | 102
Weight (lb) [Mean (Standard Deviation); unit: pounds] | 191.5 (45.2) | 171.6 (36.4) | 184.1 (31.6) | 183.8 (35.2)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Body Weight (Pounds) Change
Description: Mean percent body weight (pounds) change from baseline to 6 months post-intervention (12 months post-initiation of the intervention). Participant weight (without shoes) was measured in light clothing to the nearest 0.5 lb using a calibrated digital scale.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: percent weight change
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
percent weight change | 0.88 (3.99) | 0.53 (3.81) | -1.06 (4.37)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.1013, general linear model — The p-value above reflects results of between-arms analysis of percent change in weight from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

2. Secondary Outcome: Change in Mean HbA1c (%)
Description: Change in mean HbA1c (NGSP %) from baseline to 6 months post-intervention (12 months post-initiation of the intervention). A Siemens analyzer (point of care) was utilized to calculate HbA1c levels for each participant.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Glycated Hemoglobin
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
Percent Glycated Hemoglobin | 0.12 (1.19) | -0.30 (1.19) | 0.16 (1.01)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.4950, general linear model — The p-value above reflects results of between-arms analysis of change in mean HbA1c from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment

3. Secondary Outcome: Change in Mean Systolic Blood Pressure (mmHg)
Description: Change in mean systolic blood pressure (mmHg) from baseline to 6 months post-intervention (12 months post-initiation of the intervention). Blood pressure was measured with a sphygmomanometer, with participants seated.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
mmHg | -7.23 (12.31) | -10.71 (10.72) | -13.62 (22.5)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.7416, general linear model — The p-value above reflects results of between-arms analysis of change in systolic blood pressure from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

4. Secondary Outcome: Change in Mean Diastolic Blood Pressure (mmHg)
Description: Change in mean diastolic blood pressure (mmHg) from baseline to 6 months post-intervention (12 months post-initiation of the intervention). Blood pressure was measured with a sphygmomanometer, with participants seated.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
mmHg | 2.69 (11.69) | 0.43 (9.50) | -5.18 (15.67)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.0702, general linear model — The p-value above reflects results of between-arms analysis of change in diastolic blood pressure from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

5. Secondary Outcome: Change in Eating Habits Self-Efficacy
Description: Change in eating habits self-efficacy from baseline to 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' self-efficacy related to their ability to make healthy eating decisions in the face of real or perceived barriers (e.g. while at social events, while watching TV, etc.). This 7-item measure was adapted from items in the original Weight Efficacy Life-Style Questionnaire by Clark et al (1991) (reference provided in the References in the Protocol Section). Each of the 7 items are measured via 3 response options ("Yes/Completely Sure"=2; "Maybe/Not Sure"=1; and "No/Not Sure at All"=0), giving a possible range of scores of 0-14, with higher scores indicating higher self-efficacy for making healthy eating decisions in spite of barriers.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
scores on a scale | -0.15 (2.51) | -1.29 (3.15) | 1.76 (2.88)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.0070, general linear model — The p-value above reflects results of between-arms analysis of change in eating habits self-efficacy scores from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

6. Secondary Outcome: Change in Physical Activity Self-Efficacy
Description: Change in physical activity self-efficacy from baseline to 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' self-efficacy for exercising in the face of real or perceived barriers (e.g., bad weather, exercising alone, etc.). This 9-item measure was adapted from the Self-Efficacy for Exercise Scale by Resnick & Jenkins (2000) and Resnick et al (2004) (references provided in the References in the Protocol Section). Each of the 9 items are measured via 3 response options ("Yes/Completely Sure"=2; "Maybe/Not Sure"=1; and "No/Not Sure at All"=0), giving a possible range of scores of 0-18, with higher scores indicating higher self-efficacy for exercising despite barriers.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
scores on a scale | -0.44 (0.76) | -0.38 (0.61) | 0.28 (0.58)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.0009, general linear model — The p-value above reflects results of between-arms analysis of change in physical activity self-efficacy scale scores from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

7. Secondary Outcome: Change in Percentage of Participants Engaging in Sufficient Levels of Physical Activity Over the Past Month
Description: Change in percentage of participants engaging in sufficient levels of physical activity (PA) from baseline to 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' frequency of engaging in both moderate and vigorous levels of physical activity over the past month with two items. Both items used a 4-point response scale: 1) Rarely or Never; 2) Once a week; 3) 2-4 times a week; and 4) More than 4 times a week. Each 4-point scale for moderate PA and vigorous PA was weighted: 0=Rarely or Never; 1=Once a week; 2=2-4 times a week; and 4=More than 4 times a week. The weights were then summed and dichotomized as follows: ≥4 = sufficient PA and <4 = insufficient PA. Items were adapted to include relevant cultural examples of physical activity from the DASH 2 Brief Physical Activity Questionnaire (link to original items provided in the References in the Protocol Section).
Time Frame: Baseline, 6 months post-intervention
Population: Number of participants engaging in sufficient physical activity at baseline and 6 months post-intervention (12 months post-initiation of the intervention).
Measure: Count of Participants; unit: Participants
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 19 | 14 | 69
Participants
  Baseline | 12 | 10 | 41
  6 months post-intervention: number analyzed (Participants) | 13 | 7 | 55
  6 months post-intervention | 9 | 5 | 38
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.3740, Regression, Logistic — The p-value above reflects results of between-arms analysis for the probability of participants to engage in sufficient physical activity at 6 months post-intervention; Model adjusted for age, sex, education, marital status, employment status, and baseline physical activity

8. Secondary Outcome: Change in Sugar-Sweetened Beverage Consumption
Description: Change in participants' sugar-sweetened beverage consumption from baseline to 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' sugar-sweetened beverage consumption over the past 30 days using two questions from 'Module 14: Sugar Sweetened Beverages' of the CDC's Behavioral Risk Factor Surveillance System (BRFSS). Participants could respond in number of times per day, per week, or per month. Responses for each question were converted to number of times per day (i.e., self-reported times per week divided by 7 or self-reported times per month divided by 30), resulting in two measures: number times soda was consumed per day and number of times sugar-sweetened fruit drinks, sweet tea, and sports drinks were consumed per day. Per BRFSS guidelines, these two measures were added together to create a total daily SSB consumption rate.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: SSBs consumed per day
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 6 | 55
SSBs consumed per day | -0.71 (2.07) | -0.74 (1.52) | -0.73 (1.97)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.9556, general linear model — The p-value above reflects results of between-arms analysis of change in participants' sugar-sweetened beverage consumption per day from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

9. Secondary Outcome: Change in Fruit and Vegetable Consumption
Description: Change in participants' fruit and vegetable consumption from baseline to 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure assessed participants' fruit and vegetable consumption over the past three months using three questions adapted from: Shannon et al (1997) (reference provided in the References in the Protocol Section). Each of the three items was scored as Often=2; Sometimes=1; Never=0. Items were summed to create a scale score, giving a possible range of scores of 0-6, with higher scores indicating more frequent consumption of fruit and vegetables.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
scores on a scale | -0.38 (0.77) | 0.71 (2.14) | -0.47 (2.03)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.1726, general linear model — The p-value above reflects results of between-arms analysis of change in participants' fruit and vegetable consumption scale scores from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

10. Secondary Outcome: Change in Perceived Family Support for Exercise and Dietary Habits
Description: Change in perceived family support for exercise and dietary habits from baseline to 6 months post-intervention (12 months post-initiation of the intervention). This self-report measure was adapted to examine changes in perceived family support for engaging in healthy exercise and dietary habits. This measure consists of a 6-item scale adapted from: Gruber (2008) (reference provided in the References in the Protocol Section). Each of the 6 items are measured via 3 response options ("Often"=2; "Sometimes"=1; and "Never"=0), giving a possible range of scores of 0-12, with higher scores indicating higher perceived family support for exercising and eating healthier.
Time Frame: Baseline, 6 months post-intervention
Population: Only those with available baseline and follow-up data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | HBHS | HBHS Policy | WORD DPP
Number analyzed (Participants) | 13 | 7 | 55
scores on a scale | -0.06 (0.45) | 0.25 (0.94) | 0.48 (0.66)
Statistical Analysis 1: Comparison: HBHS vs HBHS Policy vs WORD DPP; Test type: Superiority; p = 0.0478, general linear model — The p-value above reflects results of between-arms analysis of change in participants' family support scale scores from baseline to 6 months post-intervention; Model adjusted for age, sex, education, marital status, and employment status

ADVERSE EVENTS:
Time Frame: From enrollment to 6 months post-intervention (12 months post-initiation of the study)
Description: Study staff assessed presence of adverse events via regular contact with participants from both study arms throughout the duration of the study.
Arm/Group | HBHS | HBHS Policy | WORD DPP
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/14 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14 | 0/69
Other Adverse Events (participants affected / at risk) | 0/19 | 0/14 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03377244/Prot_SAP_000.pdf